CLINICAL TRIAL: NCT03737552
Title: Sleep Patterns in Children and Adolescents With ADHD: Impact on Cognitive Functions and Quality of Life
Brief Title: Sleep Patterns in Children and Adolescents With ADHD
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mustafa M. Hashem, Principal investigator, Assiut University
Other Study IDs: SPINCD
Record Dates: First submitted 2018-11-02; First posted 2018-11-09 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Sleep Disorder; ADHD; Cognitive Change
Keywords: Sleep; ADHD; Children; Cognition
MeSH Terms: conditions — Sleep Wake Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children and adolescents with ADHD: Children and Adolescents with ADHD children or Adolescents, male or female, ages 6-17, confirmed diagnosis of Attention Deficit Hyperactivity Disorder (inattentive, hyperactive/impulsive, or combined presentations), medically healthy, no comorbid psychiatric diagnosis other than ODD, intelligence within normal limits. Participants will complete 1 night of polysomnography at sleep lab and a neuropsychological and quality of life assessment in the lab.
  Interventions: Other: Polysomnography
- Healthy control children and adolescent: children or Adolescents, male or female, ages 6-17,medically healthy, no psychiatric diagnoses, intelligence within normal limits. Participants will complete 1 night of polysomnography at sleep lab and a neuropsychological and quality of life assessment in the lab.
  Interventions: Other: Polysomnography

INTERVENTIONS:
Other: Polysomnography — Polysomnography Is considered as the gold standard of sleep assessment. It combines a number of measures of body function during sleep, including measurement of brain activity(electroencephalography),eye movements(electrooculography ),muscle activity (electromyography),heart rhythm(electrocardiography).
  Other Names: The Children's Sleep Habits Questionnaire (CSHQ); Pediatric Quality of Life Inventory 4.0 generic version; Conners' continuous performance test

SUMMARY:
This study is aimed to find out Sleep profile differences in children and adolescents with and without ADHD,Relationship between sleep profile disturbance and ADHD symptoms, Impact of sleep disturbance on cognition functions and quality of life.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is the most common neurodevelopmental disorder of childhood, affecting 3 -5% children & adolescent worldwide . Inattention, hyperactivity, and impulsiveness are the major ADHD symptoms based on the diagnostic criteria of Diagnostic and Statistical Manual of Mental Disorders (DSM), Fifth Edition .

Sleep has been referred to as a "window to the central nervous system", owing to its close associations with many other neurophysiological variables. Children are highly vulnerable to sleep disruptions in early childhood, perhaps due to the complexity of the sleep process and children's reliance on caregivers for achieving and maintaining sleep .

The relationship between sleep and ADHD is a complex process and has gained renewed interest since clinicians and researchers observed that sleep-related problems and complaints are relatively common among children with ADHD .Previous studies have shown that About 25-50% of children and adolescents with ADHD have sleep disorders , including nocturnal awakenings, phase delay, increased night time activity and insomnia.

Evaluation of sleep problems in child &adolescent clinical settings is commonly lacking, often unrecognized and go untreated in clinical setting. So, Untreated sleep disturbances and sleep disorders pose significant adverse daytime consequences and place children at considerable risk for poor health outcomes . Sleep disturbances impair a child's cognitive functioning and contribute to problems with school attendance and performance .

ELIGIBILITY:
Inclusion Criteria:

* Ages 6-17 years inclusive
* males or females
* Intelligence Quotient( IQ) > or equal 80 detected by Wechsler Intelligence Scale for Children .
* Willingness to comply with all study requirements

Inclusion criteria for ADHD group only:

• confirmed newly diagnosed ADHD according to DSM-5 Criteria. (American Psychiatric Association)

Exclusion Criteria:

* History of chronic/significant medical condition
* History or Current prescribed use of any psychotropics, including non-stimulant medications for ADHD.
* History or Current substance abuse or dependence.
* First degree relative with psychosis or bipolar disorder.

Exclusion for the ADHD group only:

• Meets criteria for any other psychiatric comorbidity Disorder besides ADHD or Oppositional Defiant Disorder (ODD).

Exclusion for the Healthy Control group only:

• Meets criteria for any psychiatric Disorders.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will involve recruitment of 51 children and adolescents with ADHD and a control group of 51 healthy childern and adolescents without psychiatric diagnoses. Participants will participate in 3 stages : Screening stage , Sleep Study stage , and Neurocognitive and quality of life assessment stage . To ensure consistency in sleep schedules, 1 night of the sleep study will occur on weeknights during the school year. The neurocognitive and quality of life assessment will occur during the afternoon following the final night of sleep assessment.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
polysomnography to measure total sleep time(minutes) in ADHD patients | 1 night
polysomnography to measure sleep efficiency(%) in ADHD patients | 1 night

SECONDARY OUTCOMES:
Assessment of cognitive function in children and adolescents with Attention Deficit Hyperactivity Disorders | 2 hours
  Conners' continuous performance test to assess cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Assad, Doctorate, Study Chair — Ain Shams University
Locations (1):
- Assiut, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lucas I, Mulraney M, Sciberras E. Sleep problems and daytime sleepiness in children with ADHD: Associations with social, emotional, and behavioral functioning at school, a cross-sectional study. Behav Sleep Med. 2019 Jul-Aug;17(4):411-422. doi: 10.1080/15402002.2017.1376207. Epub 2017 Oct 13. PMID 28922019
- [Result] Zulauf Logoz M. [The Revision and 5th Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5): Consequences for the Diagnostic Work with Children and Adolescents]. Prax Kinderpsychol Kinderpsychiatr. 2014;63(7):562-76. doi: 10.13109/prkk.2014.63.7.562. German. PMID 25478714
- [Result] Cao H, Yan S, Gu C, Wang S, Ni L, Tao H, Shao T, Xu Y, Tao F. Prevalence of attention-deficit/hyperactivity disorder symptoms and their associations with sleep schedules and sleep-related problems among preschoolers in mainland China. BMC Pediatr. 2018 Feb 19;18(1):70. doi: 10.1186/s12887-018-1022-1. PMID 29458356
- [Result] Kalil Neto F, Nunes ML. Evaluation of sleep organization in patients with attention deficit hyperactivity disorder (ADHD) and ADHD as a comorbidity of epilepsy. Sleep Med. 2017 May;33:91-96. doi: 10.1016/j.sleep.2016.08.013. Epub 2016 Oct 22. PMID 28449914
- [Result] Gad GI, Taha GR. Detection of sleep disturbances in a sample of Egyptian children attending a pediatric outpatient clinic. Middle East Current Psychiatry. 2014;21(3):185-92.
- [Result] Wechsler D. Wechsler intelligence scale for children. 1949.
- [Result] Ibrahim M, Bishry Z, Khaleel A, Ghanem M, Sheehan D, Sheehan K. Comparison of the MINI-kid with K-SADS-PL for school aged children in an Egyptian sample presented with childhood disorders [MD thesis]. Institute of Psychiatry, Ain Shams University Library. 2002.
- [Result] Asaad T KO. The Children's Sleep Habits Questionnaire. Psychometric sleep assessment instruments (Arabic version). Cairo: Center Of Psychiatry,Ain Shams University. 2001:11-3.
- [Result] El-Beh K, Hossam Eddin Khalifa H, Hassaan S, Noomani M. Measuring health-related quality of life in children with chronic medical conditions: reliability and validity of the Arabic version of PedsQL 4.0 Generic Core Scales. Middle East Current Psychiatry. 2018;25(1):16-22.
- [Result] Conners CK, Staff M, Connelly V, Campbell S, MacLean M, Barnes J. Conners' continuous performance Test II (CPT II v. 5). Multi-Health Syst Inc. 2000;29:175-96.